CLINICAL TRIAL: NCT06202261
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety and Efficacy of TQB2930 for Injection Monotherapy or in Combination for the Treatment of Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Recurrent / Metastatic Breast Cancer
Brief Title: A Study of TQB2930 for Injection Monotherapy or Combination Therapy in Patients With Recurrent/Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2930-Ib/II-01
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Breast Cancer; Recurrent Breast Cancer; Advanced Malignancies
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; Paclitaxel; Fulvestrant; Capecitabine; Vinorelbine; eribulin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TQB2930 for injection (Experimental): TQB2930 for injection,10 mg/kg, quaque week (QW), 21 day as a treatment cycle; TQB2930 for injection, 20 mg/kg, quaque 2 weeks (Q2W), 28 day as a treatment cycle; TQB2930 for injection,30 mg/kg, quaque 3 weeks (Q3W), 21 day as a treatment cycle.
  Interventions: Drug: TQB2930 for injection
- TQB2930 for injection 30mg/kg + Paclitaxel for injection (albumin-bound) (Experimental): TQB2930 for injection 30mg/kg combined with paclitaxel (albumin-bound) for injection, 21 days for one treatment cycle
  Interventions: Drug: TQB2930 for injection; Drug: Paclitaxel for injection (albumin-bound)
- TQB2930 for injection+TQB3616 capsule for injection + fulvestrant injection (Experimental): TQB2930 for injection 20mg/kg combined with TQB3616 capsule 120mg or 150mg or 180mg, and fulvestrant injection. Q2W, 28 days a cycle.
  Interventions: Drug: TQB2930 for injection; Drug: TQB3616 capsule; Drug: Fulvestrant injection
- TQB2930 for injection + chemotherapy (Experimental): TQB2930 for injection 30mg/kg combined with capecitabine tablets or vinorelbine tartrate injection or eribulin mesylate injection or gemcitabine hydrochloride for injection, 21 days a cycle.
  Interventions: Drug: TQB2930 for injection; Drug: Capecitabine tablets; Drug: Vinorelbine tartrate injection; Drug: Eribulin mesylate injection; Drug: gemcitabine hydrochloride for injection

INTERVENTIONS:
Drug: TQB2930 for injection — TQB2930 for injection is a HER2 bispecific antibody.
Drug: Paclitaxel for injection (albumin-bound) — It is an anti-microtubule chemotherapy drug
  Arms: TQB2930 for injection 30mg/kg + Paclitaxel for injection (albumin-bound)
Drug: TQB3616 capsule — TQB3616 capsule is a Cyclin-dependent kinase 4/6 (CDK4/6) inhibitor.
  Arms: TQB2930 for injection+TQB3616 capsule for injection + fulvestrant injection
Drug: Fulvestrant injection — Fulvestrant is a competitive estrogen receptor antagonist with similar affinity to estradiol
  Arms: TQB2930 for injection+TQB3616 capsule for injection + fulvestrant injection
Drug: Capecitabine tablets — Capecitabine is converted to 5-fluorouracil (5-FU) by in vivo enzyme action.
  Arms: TQB2930 for injection + chemotherapy
Drug: Vinorelbine tartrate injection — Vinorelbine is an anti-tumor drug of vinca alkaloids.
  Arms: TQB2930 for injection + chemotherapy
Drug: Eribulin mesylate injection — Eribulin induces G2/M phase cell cycle arrest, mitotic spindle division, and ultimately apoptosis after prolonged mitotic arrest through its tubulin-based anti-mitotic mechanism.
  Arms: TQB2930 for injection + chemotherapy
Drug: gemcitabine hydrochloride for injection — Gemcitabine is a cell cycle specific anti-metabolic anticancer agent
  Arms: TQB2930 for injection + chemotherapy

SUMMARY:
This is a phase Ib/II exploratory study. Phase Ib includes the dose escalation and expansion study of monotherapy, as well as the dose escalation study of combination therapy. After determining the maximum tolerated dose (MTD), a dose expansion study is conducted to observe the safety and efficacy in monotherapy. Phase II study is to further observe the safety and efficacy of TQB2930 combined with albumin-paclitaxel (cohort 3), or chemotherapy selected by investigators (cohort 4).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old; Eastern Cooperative Oncology Group Performance Status (ECOG PS) score: 0~1; The expected survival is over 3 months.
* Phase Ib

  1. Advanced malignancies confirmed by cytology / histopathology, priority given to subjects with HER2 expression or amplification;
  2. Subjects with malignant tumors who have failed standard treatment or lack effective treatment;
  3. Confirmed presence of at least one evaluable lesion according to RECIST 1.1 criteria
* Phase II

  1. Hormone receptor (HR)-negative, HER2-positive breast cancer confirmed by cytology / histopathology, with evidence of local recurrence or distant metastasis, unsuitable for surgery or radiotherapy for curative purposes:
  2. Have not received systemic antitumor therapy for metastatic stage; Systemic use of endocrine therapy is permitted, but not exceed 2 lines;
  3. at least one measurable lesion that meets the RECIST 1.1 criteria.
* Major organs are functioning normally.
* Female subjects of reproductive age should agree to use contraceptive methods during the study period and until 6 months after the end of the study; Negative serum pregnancy / urine pregnancy test within 7 days prior to study enrollment and must be non-lactating subjects; Male subjects should agree to use contraception during the study and until six months after the end of the study.

Exclusion Criteria:

* Have occured other malignant tumors within 3 years prior to first dose.
* Unalleviated toxicity above Common Terminology Criteria for Adverse Events (CTCAE) grade 1 due to any prior treatment;
* Received major surgical treatment, open biopsy, or significant traumatic injury within 28 days prior to the first dose;
* Long-term unhealed wounds or fractures;
* Arterial/venous thrombosis events occurred within 6 months before the first dose;
* Have a history of psychotropic drug abuse and can't get rid of it or have mental disorders;
* Subject with any severe and/or uncontrolled disease;
* Subjects who have been treated with other antitumor agents such as chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to the first dose, within 5 half-lives of the drug;
* Have used traditional chinese medicine with anti-tumor indications approved by National Medical Products Administration (NMPA) within 2 weeks before the first dose;
* Severe bone injury due to bone metastasis;
* Subjects with untreated active brain metastases or meningeal metastases or cancerous meningitis;
* In the course of previous HER2-targeted therapy, Left Ventricular Ejection Fractions (LVEF) decreased to <50% or absolute LVEF decreased >15%;
* Cumulative doses of anthracyclines exceeded doxorubicin or doxorubicin liposomes >360 mg/m2;
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requires continued bisphosphonate therapy
* Patients with severe hypersensitivity after the use of monoclonal antibodies;
* Has participated in other antitumor clinical trials within 4 weeks prior to the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 4 months
  The highest dose when dose-limiting toxicity (DLT) occurs in less than 33% of subjects.
Phase II recommended dose (P2RD) | Baseline up to 1 year
  Optimal tolerated dose determined after the end of phase 1
Investigators assessed Objective remission rate (ORR) based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 | Baseline up to 2 year
  The proportion of subjects with complete response (CR) and partial response (PR) whose tumor volume reduced to a predetermined value and maintained the minimum time limit.

SECONDARY OUTCOMES:
Immunogenicity | Pre-dose on Cycle 1 Day 1, Cycle 2 Day 1, Cycle 4 Day 1, Cycle 7 Day 1, Cycle 12 Day 1, each cycle is 21 or 28 days.
  Incidence of anti-drug antibody (ADA)
Peak concentration (Cmax), QW | Pre-dose, 30 minuets, 4, 8, 24, 48, 72 hours after dose on Cycle 1 Day 1, Cycle 2 Day 1; Pre-dose on Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 8, each cycle is 21 days.
  The maximum serum concentration after administration
Peak concentration (Cmax), Q2W | Pre-dose, 30 minuets, 4, 8, 24, 48, 72, 168, 240 hours after dose on Cycle 1 Day 1, Cycle 2 Day 1; Pre-dose on Cycle 1 Day 15, Cycle 2 Day 15, each cycle is 28 days.
  The maximum serum concentration after administration
Peak concentration (Cmax), Q3W | Pre-dose, 30 minuets, 4, 8, 24, 48, 72, 168, 240, 336 hours after dose on Cycle 1 Day 1, Cycle 2 Day 1; Pre-dose on Cycle 3 Day 1, each cycle is 21 days.
  The maximum serum concentration after administration
Overall survival (OS) | Baseline up to 4 years
  From randomization to the time of death from any cause.
Adverse event rate | Baseline up to 2 years
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Progression-free survival (PFS) | Baseline up to 1 year
  The time between the first medication and disease progression (PD) or death before PD.
Disease control rate (DCR) | Baseline up to 2 years
  The ratio of disease control cases (partial remission, complete response, stable disease) to total cases.
Duration of remission (DOR) | Baseline up to 2 years
  The time from the first evaluation of the tumor as a complete or partial response to the first evaluation as tumor progression or death.
Clinical benefit rate (CBR) | Baseline up to 2 years
  The ratio of disease control cases (partial remission, complete response, stable disease ≥ 6 month) to total cases.
Peak concentration (Cmax), arm 2 | Pre-dose, 30 minuets after dose of Cycle 1 Day 1,Cycle 2 Day 1, Cycle 4 Day 1,Cycle 7 Day 1,Cycle 12 Day 1,Cycle 17 Day 1. each cycle is 28 days.
  The maximum serum concentration after administration in arm 2
Peak concentration (Cmax), arm 3 and 4 | Pre-dose, 30 minuets after dose of Cycle 1 Day 1,Cycle 2 Day 1, Cycle 4 Day 1,Cycle 7 Day 1,Cycle 12 Day 1,Cycle 17 Day 1. each cycle is 21 days.
  The maximum serum concentration after administration in arm 3 and 4.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality
  - Affiliated cancer hospital of harbin medical university, Harbin, Heilongjiang